CLINICAL TRIAL: NCT05161351
Title: Evaluating the Safety of Acute Baclofen in Methadone-maintained Individuals With Opiate Dependence. An Adaptive, Single-blind, Placebo-controlled Ascending Dose Study of Acute Baclofen on Safety Parameters in Opioid Dependence During Methadone-maintenance Treatment; a Pharmacokinetic-pharmacodynamic Study
Brief Title: Evaluating the Safety of Acute Baclofen in Methadone-maintained Individuals With Opiate Dependence.
Acronym: FORWARDS-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21HH6830
Record Dates: First submitted 2021-11-04; First posted 2021-12-17 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Addiction Opiate
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Baclofen; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Adaptive, ascending-dose, parallel groups design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baclofen (Experimental): Participants will receive a single dose of either 10mg, 30mg, 60mg or 90mg of Baclofen administered as oral tablets.
  Interventions: Drug: Baclofen
- Vitamin D3 (Placebo Comparator): Participants will receive a single dose of either 20μg, 60μg or 120μg of Vitamin D3 administered as oral tablets.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Baclofen — Baclofen is the only selective GABA-B agonist licensed for human use. Originally developed as a potential anti-epileptic in the 1920s, it was found to have anti-spastic effects and is currently used for the treatment of spastic movement, especially in instances of spinal cord injury, spastic diplegia, multiple sclerosis, and amyotrophic lateral sclerosis.
  Arms: Baclofen
Drug: Vitamin D3 — Placebo tablets will be vitamin D3, (colecalciferol).
  Other Names: Placebo
  Arms: Vitamin D3

SUMMARY:
Opiate addiction is a major health challenge. The mainstay of treatment is opiate substitution therapy (OST), typically methadone, but many desire to be opiate-free. Abstinence in older opiate addicts with increasingly complex health needs may also be advantageous. Detoxification generally involves tapering of OST with adjunct medication to treat emerging symptoms, but these are often ineffective or inappropriate for longer-term prescribing. New treatments are therefore needed. The investigators propose that baclofen has the desired properties to facilitate OST detoxification. It is licensed for spasticity, is currently used to treat alcoholism and there is promising pre-clinical and clinical evidence of potential efficacy in opiate dependence. Common symptoms of withdrawal are likely to be improved by baclofen. Whilst the investigators clinical experience and other studies suggest baclofen can be taken safely with methadone, they could potentially interact causing adverse effects such as respiratory depression. Also, the possibility of abuse liability remains unexplored and is an important consideration in this indication. The investigators will therefore determine the safe dose combinations of baclofen and methadone and to assess if baclofen is 'liked'. Patients engaged in treatment for opiate dependence from community addiction services and receiving stable doses of OST with methadone will be invited to undergo screening at the Imperial Clinical Research Facility (ICRF) at Hammersmith hospital, or at their local addiction clinic. Up to 64 eligible patients will attend the ICRF for an experimental visit. Acute baclofen or placebo will be orally administered (randomised, single-blind, 3:1 ratio respectively) with the dose determined by a Bayesian adaptive trial algorithm. Measures will comprise respiratory, sedation, self-report and cardiovascular monitoring, and blood sampling for 5 hours post-dose. The study duration will be ~2-3 weeks from pre-screening phone call to the post visit follow up phone call.

DETAILED DESCRIPTION:
This study will evaluate the safety of acute baclofen in methadone-maintained individuals with opiate dependence. The goal of the trial is to study the safety of these drugs given in combination using an adaptive, single-blind, placebo-controlled ascending dose design investigating the impact on respiratory, cardiovascular and pharmacokinetic-pharmacodynamic (PK-PD) parameters.

This study will determine the maximum safe dose of baclofen depending on the prescribed dose of methadone. Methadone doses will vary depending on the recruited cohort, but the investigators anticipate an average dose of ~53mg (range 5 to 120mg), based on data from local drug and alcohol services. The investigators are seeking a minimum safe dose of 30mg baclofen in combination with a minimum of 60mg methadone. Findings will be used to inform a subsequent proof-of-concept trial of the efficacy of baclofen. The investigators will investigate each of the four factors of i) safety, ii) dose-response, iii) potential for abuse liability and iv) objective and subjective measures of GABA-B receptor sensitivity, providing clarity on the relationship between these factors. The investigators will include a placebo arm to evaluate the pharmacodynamic effects of baclofen, and to control for expectation effects.

Safety will be established using a Bayesian dose-escalation adaptive model which will be informed by the occurrence of dose-limiting toxicity (DLT) events at increasing doses of baclofen at the following dose levels: 10, 30, 60, 90mg. The evaluation window for all outcomes will begin at dosing and end at 5 hours post-dose, with further follow-up by phone the following day. The DLT of primary concern is respiratory depression, and the investigators consider that the risk increases with the dose of baclofen and methadone-maintenance level. Formally, the objective is to find the combination associated with 15-25% risk of a DLT. The combination-toxicity response will be evaluated using the continual reassessment method, a model-based design for trials that aim to find the maximum tolerated dose, where the baclofen dose recommendation for each given patient with prescribed dose of methadone will be supported by the adaptive Bayesian model. Participants will be randomised (single-blind) to baclofen or placebo in a 3:1 ratio. If allocated to baclofen, participants will be dosed in groups of up to 3, with a maximum sample size of 48 allocated to baclofen, and 16 to placebo.

Outcome measures that will be used to determine the incidence of a DLT will include oxygen saturation, respiratory rate, cardiovascular measures (ECG, blood pressure) and CNS effects (sedation, alertness). Transcutaneous CO2 and adverse events will also be monitored.

The adaptive Bayesian model will be regularly updated (after each group of up to 3 participants administered baclofen) given the observed patients' responses, providing efficiency in decision-making, by recommending the most likely safe target individualised dose. The study can therefore be stopped earlier for safety if the model suggests that 30mg of baclofen and 60mg of methadone is highly likely to be unsafe.

The study can also stop earlier if the highest dose of baclofen (90mg) is highly likely to be safe, i.e. shows no DLTs with 120mg of methadone, provided that the study has also achieved sufficient data to meet secondary endpoints.

In addition to the approach described above, an evaluation of pharmacokinetic parameters will be investigated through regular blood sampling and assay of baclofen and methadone plasma concentrations. The pharmacodynamic effects of baclofen relative to placebo, and their dose separation will be determined through objective (plasma growth hormone concentrations) and subjective measures (visual analogue scales and questionnaires for drug effects, anxiety, sleep). The potential for abuse liability, relative to placebo, will be assessed using the Drug Effects Questionnaire.

GABA-B receptor sensitivity will be determined through comparison of pharmacodynamic effects in comparison with historical healthy controls, using data derived from previous work using comparable measures and time-points at the 10 and 60mg baclofen dose levels.

Primary & secondary endpoints: If the investigators find that all dose levels of baclofen are safe up to and including 90mg in combination with 120mg methadone (primary endpoint), the study can still continue up to the maximum sample size to achieve maximum precision for secondary outcomes, explore more methadone doses (<120mg) in a variety of participants and baclofen dose-response separation, as required.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged over 21
3. Willing and able to comply with protocol
4. Able to read, comprehend and record information written in English
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
6. Healthy as determined by a responsible physician, based on a medical evaluation which includes medical history, a physical examination, laboratory tests (if required), and a psychiatric evaluation. A volunteer with clinical parameters outside the reference range for the population being studied may be included, only if the investigators concur that the finding is unlikely to jeopardize either subject safety or study integrity.
7. DSM-5 diagnosis of current severe opioid use disorder
8. Treated with methadone substitution therapy and able to maintain the same stable dose for screening and experimental visit.
9. Ability to receive an acute dose of up to 90mg baclofen or up to 4800IU vitamin D (placebo).

Exclusion Criteria:

1. Intoxication on any of the visits, as assessed by difficulty in walking, the slurring of speech, difficulty concentrating or drowsiness. This exclusion criteria would exclude a subject from that study day only and not the whole study, at the discretion of the research team.
2. Positive urine drug screens or breath alcohol at screening or experimental testing visits. A minimum list of drugs that will be screened for include amphetamines, cocaine, opiates, methadone, cannabinoids and benzodiazepines. Positive results for methadone will be allowed for those opiate dependent participants still undergoing OST. Positive results for cannabinoids will be allowed given the long half-life of cannabinoid metabolites. This exclusion criteria would exclude a subject from that study day only and not the whole study, at the discretion of the research team.
3. Current DSM-5 substance dependence disorder for any other substance except for opiates and nicotine. Lifetime history of dependence on other substances will be allowed given very high incidence of co-dependence.
4. Regular on-top use of heroin or other opiates or other illicit substances in combination with OST, which in the opinion of the investigators will interfere with subject safety or study integrity.
5. Any participant taking over 120mg/day of prescribed methadone.
6. Current severe DSM-5 mental health disorder (excluding opiate dependence). Current moderate or mild DSM-5 depressive, anxiety, sleep or personality disorders will be allowed given the high levels of comorbidity, provided in the opinion of the investigators, the participant is able to complete study procedures satisfactorily.
7. Current or past history of enduring severe mental illness e.g. psychotic disorder (excluding drug induced), schizophrenia, bipolar affective disorder).
8. Active suicidality.
9. Use of regular prescription medications which in the opinion of the investigators will interfere with subject safety or study integrity. Regular use of psychotropic medication will be permitted e.g. antidepressants, provided the participant is compliant with administration and the investigators concur that they will not interfere with subject safety or study integrity.
10. Participants are taking any medication that is contraindicated with baclofen or placebo (vitamin D3), or are hypersensitive to them or any of their excipients.
11. Participants that are taking any medication that in the opinion of the investigators may impact on the outcome measures during the experimental session.
12. Use of intermittent psychotropic medication which in the opinion of the investigators will interfere with subject safety or study integrity.
13. End stage or acute renal failure.
14. Severe chronic obstructive pulmonary disease (COPD) or Type 2 respiratory failure.
15. Pulse rate <40 or >100 BPM OR systolic blood pressure >160 and <100 and a diastolic blood pressure >95 and <60 in the semi-supine position.
16. Oxygen saturation <92% at rest
17. A screening ECG with a QTcB or QTcF > 500 msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave) and/or with another ECG abnormality which in the opinion of the study physician is clinically significant and represents a safety risk. Note that if the initial QTc value is prolonged, the ECG should be repeated two more times (with 5 minutes between ECG readings) and the average of the 3 QTc values used to determine eligibility.
18. Clinically significant head injury (e.g., requiring medical or surgical intervention) that in the opinion of the investigators, contraindicates their participation .
19. Active hepatitis or HIV.
20. Active peptic ulceration.
21. Significant current or past medical history that, in the opinion of the investigators, contraindicates their participation.
22. The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the first experimental visit.
23. Pregnancy or breast-feeding
24. Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare Trust, London, United Kingdom

REFERENCES:
- [Result] Paterson LM, Barker D, Cro S, Mozgunov P, Phillips R, Smith C, Nahar L, Paterson S, Lingford-Hughes AR. FORWARDS-1: an adaptive, single-blind, placebo-controlled ascending dose study of acute baclofen on safety parameters in opioid dependence during methadone-maintenance treatment-a pharmacokinetic-pharmacodynamic study. Trials. 2022 Oct 18;23(1):880. doi: 10.1186/s13063-022-06821-9. PMID 36258248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited only 16 patients in the end, as the primary outcome measure was met, and each person from the 16 patients only received one dose.
Groups:
- Period 1 Baclofen 10mg: Participants will receive a single dose of 10mg of Baclofen administered as oral tablets.
  Baclofen: Baclofen is the only selective GABA-B agonist licensed for human use. Originally developed as a potential anti-epileptic in the 1920s, it was found to have anti-spastic effects and is currently used for the treatment of spastic movement, especially in instances of spinal cord injury, spastic diplegia, multiple sclerosis, and amyotrophic lateral sclerosis.
- Vitamin D3: Participants will receive a single dose of either 20μg (to match period 1), 60μg (to match period 2) or 120μg (to match period 3) of Vitamin D3 administered as oral tablets.
  Vitamin D3: Placebo tablets will be vitamin D3, (colecalciferol).
- Period 2 Baclofen 30mg: Participants will receive a single dose of 30mg of Baclofen.
- Period 3 Baclofen 60mg: Participants will receive a single dose of 60mg of Baclofen
Period: Overall Study
Arm/Group | Period 1 Baclofen 10mg | Vitamin D3 | Period 2 Baclofen 30mg | Period 3 Baclofen 60mg
Started | 3 (14 were assigned but only 12 started baclofen) | 4 | 5 | 4
Completed | 3 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baclofen 10mg: Participants will receive a single dose of 10mg of Baclofen administered as oral tablets.
  Baclofen: Baclofen is the only selective GABA-B agonist licensed for human use. Originally developed as a potential anti-epileptic in the 1920s, it was found to have anti-spastic effects and is currently used for the treatment of spastic movement, especially in instances of spinal cord injury, spastic diplegia, multiple sclerosis, and amyotrophic lateral sclerosis.
- Baclofen 30mg: Participants will receive a single dose of 30mg of Baclofen administered as oral tablets.
- Baclofen 60mg: Participants will receive a single dose of 60mg of Baclofen administered as oral tablets.
- Total: Total of all reporting groups
Arm/Group | Baclofen 10mg | Vitamin D3 | Baclofen 30mg | Baclofen 60mg | Total
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (3.1) | 46 (7.4) | 45.8 (12.6) | 47.5 (6.4) | 46.8 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 2
  Male | 2 | 4 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 5 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 4 | 5 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: The maximum safe dose of baclofen at which 15-25% of evaluable participants experience a dose limiting toxicity (DLT) for prescribed doses of methadone
Time Frame: up to 24 hours after dosing
Measure: Number; unit: participants
Groups:
- Baclofen 30mg: Participants will receive 30mg of baclofen
- Baclofen 60mg: Participants will receive 60mg of Baclofen
Arm/Group | Baclofen 10mg | Vitamin D3 | Baclofen 30mg | Baclofen 60mg
Number analyzed (Participants) | 3 | 4 | 5 | 4
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study day and following morning.
Groups:
- Baclofen 10mg: Participants will receive a single dose of 30mg of Baclofen administered as oral tablets.
  Baclofen: Baclofen is the only selective GABA-B agonist licensed for human use. Originally developed as a potential anti-epileptic in the 1920s, it was found to have anti-spastic effects and is currently used for the treatment of spastic movement, especially in instances of spinal cord injury, spastic diplegia, multiple sclerosis, and amyotrophic lateral sclerosis.
Arm/Group | Baclofen 10mg | Vitamin D3 | Baclofen 30mg | Baclofen 60mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 2/5 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen 10mg (N=3) | Vitamin D3 (N=4) | Baclofen 30mg (N=5) | Baclofen 60mg (N=4)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT05161351/Prot_SAP_000.pdf